CLINICAL TRIAL: NCT00384462
Title: A Prospective, Non-Interventional Study to Evaluate the Incidence of Hospitalizations and Medically-Attended Lower Respiratory Tract Infection (MALRI) in Premature Infants 32 to 35 Weeks Gestational Age Who Are Not Recommended to Receive Prophylaxis for RSV
Brief Title: Study to Evaluate the Incidence of Hospitalizations and Respiratory Tract Infections in Premature Infants
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Frank Malinoski, M.D., PhD, MedImmune Inc.
Other Study IDs: MI-MA140
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Premature infants (32-35 weeks GA) <6 months of age at the start of the RSV season who are not receiving palivizumab and do not have CLD of prematurity; Respiratory Syncytial Viruses
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Premature Infants (32-35 wks. GA) who are less than six months of age at start of RSV season and followed until May of the following year.
- 2: Premature newborns (32-35 wks. GA) who are born during the current RSV season and discharged from the hospital after 01 Dec and followed until May of the next year.

SUMMARY:
The purpose of this study is to describe respiratory syncytial virus (RSV) hospitalization rates and to begin to address the utilization of outpatient resources for RSV medically-attended lower respiratory tract infections (MALRI) in 32-35 week gestational age (GA) premature infants who are less than 6 months of age and do not receive treatment.

DETAILED DESCRIPTION:
The goals of this study are:

* To estimate the incidence of hospitalization attributable to RSV within 150 days from enrollment in premature infants who are:

  * 32-35 weeks GA
  * less than 6 months of age at the start of the RSV season
  * not receiving palivizumab prophylaxis and not recommended to receive palivizumab according to the AAP guidelines
* To estimate the incidence rate of hospitalization attributable to RSV in the other relevant study populations and time periods (e.g., Cohort 2, Cohorts 1 and 2 combined, and subgroups based on chronological age at the start of the RSV season, GA, etc. within 150 days from enrollment and other time periods based on RSV activity, etc.)
* To estimate the incidence of RSV-associated MALRI in the study populations
* To characterize the incidence and type of clinical interventions for MALRI in the study populations

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian able to understand and provide written informed consent
* Male or female infants born at 32-35 weeks GA. GA will be determined according to available medical records.
* Clinically stable, in the opinion of the investigator
* Ability and willingness of the subject's parent/legal guardian to complete all protocol mandated follow-up telephone calls, visits and procedures
* Not more than one of the following American Academy of Pediatrics (AAP)-defined risk factors:

  1. Childcare attendance
  2. School-aged siblings in the home
  3. Exposure to environmental air pollutants (not including passive exposure to tobacco smoke)
  4. Congenital abnormalities of the airways
  5. Severe neuromuscular disease, as determined by the investigator
* Subject must meet the criteria listed below for either Cohort 1 or Cohort 2:

Cohort 1

* Date of enrollment between 01/Oct and 15/Dec
* Chronological age of < 6 months (i.e., has not yet reached 6-month birthday) at the traditional start of the local RSV season (as used to determine eligibility for RSV prophylaxis)

Cohort 2

* Date of enrollment between 16/Dec and 15/Feb
* Born during the current RSV season and discharged from the hospital nursery after 01/Dec

Exclusion Criteria:

* Previous (within 90 days of enrollment) or concurrent treatment with palivizumab or RSV-IGIV or IVIG
* Hospitalization at the time of enrollment (unless discharge is anticipated within 10 days)
* Two or more AAP-defined risk factors as listed under Inclusion Criteria
* Participation in trials of investigational RSV prophylaxis or therapeutic agents
* Confirmed prior or current RSV infection (a child with current signs/symptoms of respiratory infection must have negative RSV testing)
* Diagnosis of chronic lung disease (CLD) of prematurity (formerly referred to as bronchopulmonary dysplasia [BPD])
* Diagnosis of hemodynamically significant congenital heart disease (CHD), defined as requiring medication or supplemental oxygen for their CHD
* Known immunodeficiency
* Life expectancy of < 6 months

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2 cohorts of premature infants and premature newborns 32-35 weeks
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Estimate the incidence of hospitalization attributable to RSV within 150 days from enrollment in premature infants | 150 days from enrollment

SECONDARY OUTCOMES:
Estimate the incidence rate of hospitalization attributable to RSV in the other relevant study populations | 150 days after enrollment
Estimate the incidence rate of MALRI attributable to RSV in the study populations; | during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Frank Malinoski, M.D., PhD, Study Director — MedImmune LLC
Locations (59):
- United States (59):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Central Arkansas Pediatric Clinic, P.A., Benton, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Little Rock Children's Clinic, Little Rock, Arkansas
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital of Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital, Denver, Colorado
  - Pediatric Pulmonology, LLC, Stamford, Connecticut
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - University of Miami Medical Center, Miami, Florida
  - University of South Florida Pediatrics Ambulatory Care Center, Tampa, Florida
  - Georgia Pediatric Pulmonology Associates, Atlanta, Georgia
  - Kapiolani Medical Center, Honolulu, Hawaii
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Maryland, School of Medicine, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Children's Healthcare D.B.A. Hospitals & Clinics, Saint Paul, Minnesota
  - Pediatrix Medical Group, St. John's Mercy Medical Center, St Louis, Missouri
  - Midwest Children's Health Research Institute, LLC, Lincoln, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - Winthrop University Hospital, Mineola, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Hospital, State University of New York at Stony Brook, Stony Brook, New York
  - Crouse Hospital NICU, Syracuse, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Raleigh Pediatric Associates, Gardner, North Carolina
  - Raleigh Pediatric Associates, Raleigh, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Beehly Medical Park Women's and Children's Pavilion, Boardman, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - Children's Medical Center, Dayton, Ohio
  - Pediatric Associates of Dayton, Inc., Kettering, Ohio
  - St. Vincent Medical Center, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Geisinger Medical Center - JW Children's Hospital, Danville, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Houston Medical Center, Houston, Texas
  - VCU Medical Center, Children's Pavillion, Richmond, Virginia
  - University Physicians Internal Medicine, Huntington, West Virginia
  - West Virginia University, Morgantown, West Virginia
  - Children's Hospital Waukesha Memorial, Waukesha, Wisconsin
  - Children's Corporate Center, Wauwatosa, Wisconsin